CLINICAL TRIAL: NCT03431467
Title: A Prospective Randomised Trial of Early LV Venting Using Impella CP for Recovery in Patients With Cardiogenic Shock Managed With VA ECMO
Brief Title: Impella CP With VA ECMO for Cardiogenic Shock
Acronym: REVERSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael Ibrahim, Co-Principal Investogator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 828198
Record Dates: First submitted 2018-01-21; First posted 2018-02-13 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cardiogenic Shock
Keywords: ECMO; Heart Failure; RCT; Mechanical unloading
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial at three U Penn Sites
Who Masked: Outcomes Assessor
Masking Description: All data will be masked as far as possible. For example, Echo data will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): VA-ECMO alone per standard clinical protocol.
- Experimental (Experimental): VA-ECMO with early institution of Impella CP LV venting
  Interventions: Device: Impella-CP LV Vent

INTERVENTIONS:
Device: Impella-CP LV Vent — Patients randomised to the experimental arm will have an Impella-CP implanted in addition to VA-ECMO within a maximum of 10 hours of institution of VA-ECMO
  Arms: Experimental

SUMMARY:
Veno-arterial extra-corporeal membrane oxygenation (VA-ECMO) is indicated as a haemodynamic rescue strategy in decompensated acute or chronic heart failure presenting as cardiogenic shock. It has been used across aeitologies including post-myocardial infarction, dilated cardiomyopathy, acute myocarditis and in post-cardiotomy shock. VA ECMO has a number of effects on the circulation including improved end-organ perfusion and possibly improved coronary perfusion, and is a bridge to further therapies including permanent advanced mechanical circulatory support, cardiac transplantation and to cardiac recovery.

Left ventricular assist devices (LVADs) provide long-term mechanical circulatory support and also profoundly mechanically unload the left ventricle. Multiple clinical studies have documented cardiac recovery using LVAD therapy, with a rate between 10-60% in selected populations. A large body of basic science has documented the pivotal role of mechanical load in determining ventricular contractile performance across species. Therefore both clinical data and basic laboratory studies support the notion that profound ventricular unloading may result in improved cardiac performance through a variety of mechanisms ranging from triggered de novo cardiomyocyte proliferation, subcellular calcium handling reverse remodeling, changes to the extracellular matrix of the heart, reverse remodeling of the neurohormal milleu, amongst many others.

One of the major deficiencies of peripheral VA-ECMO is its lack of left ventricular unloading, with associated pulmonary congestion, which can derail clinical improvement and hamper cardiac recovery. Indeed, percutaneous VA-ECMO increases LV afterload due to the retrograde blood flow, and because of the lack of venting, there may be progressive LV distension. These conditions can result in a congested, pressure-overloaded ventricle, even in the absence of echocardiographic ventricular distension. This may be ameliorated with the addition of ventricular mechanical unloading using percutaneous therapies including the percutaneous left ventricular device, Impella CP.

On the platform of VA-ECMO, the addition of an Impella device to reduce ventricular loading results in improved survival and recovery of ventricular performance in the setting of cardiogenic shock. In a number of small studies, the use of additional means to unload the ventricle, principally Impella, results in cardiac recovery and less ventricular distension. In chronic heart failure, direct ventricular unloading is critical to cardiac recovery.

The objective of this randomized study is to determine whether the addition of early direct ventricular unloading using Impella CP leads to higher rates of cardiac recovery, defined as survival free from mechanical circulatory support, heart transplantation or inotropic support at thirty days. This study will also examine the clinical, biochemical, echocardiographic and radiologic effects of VA ECMO with and without the addition of Impella CP to directly vent the left ventricle to address adjunct important questions such as the effects on pulmonary congestion.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock: Including refractory to conventional therapy, including systolic blood pressure < 90mm Hg, Cardiac Index < 1.8 or a cardiac index < 2.0 on moderate to high doses of inotropes and vasopressors for greater than 30 mins, or systemic signs of tissue hypoxia.
* Post-acute myocardial infarction cardiogenic shock: excluding mechanical complications requiring surgical intervention after extracorpeal membrane oxygenator (ECMO) such as post-ischaemic ventricular septal defect (VSD).
* Drug overdose-induced cardiogenic shock.
* Early graft failure: post orthotropic heart transplantation cardiogenic shock, excluding immediate intra-operative failure.
* Acute on chronic cardiomyopathy with progressive shock and decompensation unresponsive to medical therapies.

Exclusion Criteria:

* Recent Significant Pulmonary Embolus
* Moderate to severe aortic valve insufficiency (AI)
* Ongoing significant sepsis
* Severe pulmonary hypertension & shock
* Hypothermia
* Post-cardiotomy cardiogenic shock
* Continuous cardiopulmonary resuscitation (CPR) >20-30 minutes, except if neurological status is satisfactory
* Transfer from outside hospital on VA ECMO or with history of CPR
* Listed for cardiopulmonary transplantation or being evaluated for cardiopulmonary transplantation or permanent mechanical circulatory support
* Known or suspected chronic heart failure with echocardiogram documenting left ventricular diastolic diameter >6.5cm
* Known or suspected chronic heart failure with echocardiogram documenting left ventricular ejection fraction < 25%
* Mechanical aortic valve replacement
* Presence of left ventricular thrombus
* Pre-existing Impella 2.5, CP, 3.5 or 5.0
* Cardiogenic shock due to primary respiratory failure
* Mechanical complications requiring surgical intervention after ECMO such as post-ischaemic VSD.
* Severe liver failure
* Active malignancy
* Acute aortic dissection
* Intracranial hemorrhage
* Neurological injury including recent cerebrovascular accident or suspected severe neurologic injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Bermudez, MD, Principal Investigator — University of Pennsylvania; Michael Ibrahim, MD PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Deidentiifed data will be used within the research team

REFERENCES:
- [Derived] Moussa MD, Roux J, Jungling M, Ramdane N, Loobuyck V, Brassart B, Rousse N, Dupre C, Mugnier A, Khalipha A, Bardeesi ASA, Lukowiak O, Lefebvre L, Juthier F, Robin E, Labreuche J, Thellier L, Vincentelli A. Impella Versus Selective Biatrial Canulation for Left Ventricular Unloading During Extracorporeal Membrane Oxygenation. Cardiovasc Ther. 2026 Feb 8;2026:3669575. doi: 10.1155/cdr/3669575. eCollection 2026. PMID 41668891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Recovery From Cardiogenic Shock.
Description: The number of subjects treated with this standardized ECMO protocol with either (i) no additional therapy or (ii) Impella CP for LV mechanical unloading who experience myocardial recovery defined as: survival free from mechanical circulatory support, heart transplantation or inotropic support.
Time Frame: At forty five days.
Population: Survival free from mechanical circulatory support, heart transplantation or inotropic support at 40 days.
Measure: Count of Participants; unit: Participants
Groups:
- Control 40 day Survival: VA-ECMO alone per standard clinical protocol survival at 40 days.
- Experimental 40 Day Survival: VA-ECMO with early institution of Impella CP LV venting survival at 40 days.
  Impella-CP LV Vent: Patients randomised to the experimental arm will have an Impella-CP implanted in addition to VA-ECMO within a maximum of 10 hours of institution of VA-ECMO
Arm/Group | Control 40 day Survival | Experimental 40 Day Survival
Number analyzed (Participants) | 9 | 8
Participants
  Survival at Discharge | 5 | 4
  In Hospital Mortality | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment through removal of ECMO and at hospital discharge, 30 days (+/-15 days) and 180 days (+/- 60 days) after initial ECMO institution.
Description: Serious Adverse Events (SAEs) and any unexpected SAEs will be collected from the time of ECMO insertion through removal and hospital discharge. All SAEs will be reported using modified INTERMACS adverse event (AE) categories. The INTERMACS AE definitions have been modified to exclude pediatrics and include SAEs related to extracorporeal mechanical assist devices, including percutaneous cannula insertion.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 4/8 | 4/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=8) | Experimental (N=8)
Loss of pulse (Vascular disorders) | 2 | 0
Thromboembolism (Vascular disorders) | 3 | 2
Localized non-device infection (Infections and infestations) | 2 | 0
Percutaneous cannula site infection (Infections and infestations) | 1 | 0
Cardiac arrythmias (Cardiac disorders) | 1 | 2
Neurological dysfunction (Nervous system disorders) | 1 | 2
Major bleeding (Vascular disorders) | 1 | 0
Washout (Surgical and medical procedures) | 1 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 0
Renal dysfunction (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
1. Difficulty in enrollment due to the perception of needing infrequent unloading and/or that unloading was not necessary.
2. Impella 5.5 was released during the trial. Impella 5.5 was. more potent that the Impella CP.
3. COVID-19 pandemic restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03431467/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03431467/SAP_001.pdf